CLINICAL TRIAL: NCT05305209
Title: Efficacy of K-laser as a Therapeutic Treatment of the Symptoms of Genitourinary Syndrome of Menopause (SGM) in Postmenopausal Women: a Randomized Clinical Trial
Brief Title: Laser Therapy for Treatment of Genitourinary Syndrome of Menopause (GSM) in Postmenopausal Women
Acronym: LASER_2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Collaborators: Antonia Maria Ruiz Moreno (Unknown); María Dolores Martínez Colmena (Unknown); María del Carmen Iniesta Moreno (Unknown); María Lydia Serra Llosa (Unknown)
Responsible Party: Principal Investigator, Rocío Martín Valero, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UMA _SGM_2022
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: GSM (genitourinary syndrome of menopause); laser treatment; postmenopausal condition; urinary incontinence; vulvovaginal atrophy
MeSH Terms: conditions — Urinary Incontinence | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): They will receive the k-laser treatment with the k-laser Cube Plus 30 device
  Interventions: Other: Intervention group
- Control Group (Placebo Comparator): They will receive a sham treatment with the k-laser Cube Plus 30 device turned off
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention group — The patients will receive 12 minutes of intravaginal application with an average power of 1 watios and total applied energy of 720J and an extracavitary application for 4 minutes with an average power of 3 watios and a total dose of 720J with all effects at 200%, twice a week for 6 weeks.
  Arms: Intervention group
Other: Control Group — The patients will receive 12 minutes of intravaginal application and 4 minutes of extracavitary application, twice a week for 6 weeks. The difference compared to the intervention of group 1 is that the device will be off and therefore will not emit energy.
  Arms: Control Group

SUMMARY:
This is a prospective, multi-centre, double blinded, randomized controlled trial, which will be conducted under a common protocol.

The aim of this study is to evaluate the efficacy of vaginal laser for treatment of GSM (Genitourinary Syndrome of Menopause) compared to the sham procedure in postmenopausal women.

The study population is female subjects > 18 years old with symptoms of genitourinary syndrome of menopause (GSM) who have not menstruated for at least 5 years.

DETAILED DESCRIPTION:
The clinical data will be analysed by comparing post-treatment data with the baseline data (clinical history, compliance with selection, inclusion and exclusion requirements, assessment of the muscle and pH, and questionnaires). The follow-up is for 6 weeks after the procedure, a physical examination will be passed again to assess whether the effects on the tissue are maintained once the treatment is finished (coloration, hydration, and mobility of the tissue). Two biopsies will be taken, once at the beginning of treatment and another at the end.

The symptoms of SGM worsen as the age of the subject advances, which is why a treatment is required that improves the symptoms in the long term and maintains them once the treatment is finished. For this reason, the objective is to carry out a randomized control study with a new K-Laser Cube device that minimizes the possible risks of conventional vaginal laser therapy.

The hypothesis is that women who will undergo vaginal K-Laser treatment will report an improvement not only in SGM, but also in pelvic floor dysfunctions. The objective in this pilot study will be to evaluate the effects of K-laser treatment on pelvic floor dysfunctions using validated and commonly used questionnaires.

Changes in vaginal pH measured by FSFI (Female Sexual Function Index) questionnaire and changes in the deep musculature with the PERFECT protocol and the OXFORD scale will be the primary endpoints of the study. The secondary endpoints include quality of life changes with the SF-12 (Short Form) health questionnaire and Cervantes Scale, CPPQ-Mohedo (Chronic Pelvic Pain Floor) questionnaire, PFDI-20 (Pelvic Floor Distress Inventory) questionnaire and the Menopause Rating Scale (MSR).

ELIGIBILITY:
Inclusion Criteria:

* Women of any age with established menopause of 5 years or more who report genitourinary discomfort, dyspareunia, sequelae, genital atrophy, voiding discomfort, voiding urgency or urinary incontinence. Postmenopausal status is defined if patients have at least 12 continuous months of amenorrhea for no other apparent reason or permanently elevated follicle-stimulating hormone (FSH) blood levels (≥30 mIU/mL).
* Patients who have had cancer treatment already completed and in the process of remission.
* Sexually active
* Nulliparous or who have had vaginal deliveries or caesarean section
* That they do not receive hormone replacement therapy in any of its routes of administration. If you received HRT, 4 months must have elapsed since stopping treatment before starting the trial protocol.
* Motivated and committed to complete the trial

Exclusion Criteria:

* According to the pelvic organ prolapse quantification system [POP-Q], POP>Stage 2, , severe urinary or fecal incontinence (FI) or any disease that could influence the study protocol. In addition, patients will be advised to refrain from vaginal practices for three days prior to each biopsy (one at the beginning and one at the end of treatment).
* Women who are not sexually active, do not have coital relationships, either with a partner or alone
* Women with recurrent cystitis or candidiasis
* Women with little motivation to participate in the trial
* Minors
* Patients who do not have the ability to comprehend or understand what participation in a clinical trial entail
* Patients with severe psychiatric pathology (depression, anxiety)
* Patients with degenerative neurological pathology: either cognitive impairment or ALS, MS, diabetic neuropathy, etc.
* Patients with neuropathic genital pain (neuralgia or pudendal nerve entrapment)
* Vulvodynia, hyperalgesia, or genital allodynia
* Post-pelvic surgery of less than 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Vaginal pH | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  During the physical examination a sample of the mucosa will be extracted to check the acidity of the pH. This is a marker of the health of the vaginal flora and abnormalities in pH values will be determined by hormonal imbalances of oestrogens. A pH> 4.5 refers to a decrease in local vaginal defenses which predisposes to infections or inflammatory processes. The pH analysis is a valid tool to diagnose menopause equivalent to an analysis of the levels of the follicle-stimulating molecule (FSH) non-invasive and inexpensive.
Change from Baseline in the deep musculature with the PERFECT protocol | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  Digital evaluation is essential during the examination of the pelvic floor muscles. For this, digital palpation and a pressure gauge will be used. Digital assessment is performed by inserting the index and middle fingers into the distal 3 centimetres of the vagina in a frontal plane.
  The PERFECT protocol is described as an acronym for evaluating the main components of pelvic floor muscle contractility. The components are: P (power, score muscle strength according to the OXFORD scale), E (endurance, time the maximum contraction is maintained without loss of strength), R (repetitions, number of contractions with intervals of 4 to 10 seconds), F (number of fast contractions followed after a rest of 1 minute), ECT (every contraction timed: each contraction measured) that consists in evaluating each contraction before the beginning of the treatment, which allows individualizing the program.
Analysis of the impact on QoL (Quality of life) with the FSFI (Female Sexual Function Index) questionnaire. | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  FSFI questionnaire assesses sexual function in women with pelvic floor dysfunction. It consists of 6 domains and 19 items (Cronbach's alpha coefficient =0.85). The maximum score is 36.0 (high level of sexual functional) and minimum score is 2.0 (low level of sexual functional). The domains are: desire (2 items), arousal (4 items), lubrication (4 items), orgasm (3 items), satisfaction (3 items), pain (3 items).

SECONDARY OUTCOMES:
Analysis of the impact on QoL (Quality of life) with the SF-12 (Short Form) health questionnaire. | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  This questionnaire is the reduced Spanish version of the SF-36 general health questionnaire, which has 35 items divided into 8 dimensions (physical function, physical role, emotional role, social function, mental health, general health, body pain and vitality). The SF-12 questionnaire has 12 items distributed in 2 health components: physical (CSF) with a Cronbach's alpha coefficient of 0.85 and mental (CSM) with a Cronbach's alpha coefficient of 0.78. It is one of the most widely used generic instruments for evaluating health-related quality of life.
Analysis of the impact on QoL (Quality of life) with Cervantes Scale | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  The Cervantes scale is a questionnaire to measure health-related quality of life. It is a tool specifically designed and validated for menopause in Spanish women, original in Spanish and adapted to our environment. The definitive scale consists of 31 items and 2 dimensions: menopause and health. 15 items are related to vasomotor symptomatology, health and aging; 4 items with sexuality; 3 items with the couple relationship and 9 items with psychic domain. The global Cronbach's alpha coefficient is 0.909 and that of the different subscales between 0.79 and 0.85. It is a short scale and easy and quick to apply, approximately 7 minutes. The bases fluctuate between 0 (best quality of life) and 155 (worst quality of life). Its age of application is the Spanish female population between 45 and 64 years old and it has scales to compare the results with younger women or of the same age.
Assessment of pain with the CPPQ-Mohedo (Chronic Pelvic Pain Floor) questionnaire | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  This questionnaire consists of 7 questions and is a screening tool to identify patients and include them in treatment programs, it allows the evaluation of results for treatments and clinical trials, as well as evaluating the prevalence of chronic pelvic pain in epidemiological studies. For the preparation of the CPPQ-Mohedo questionnaire, the NIH-CPSI (questionnaire for the evaluation of chronic prostatitis, male sex) was used and to test the ability to discriminate between healthy and unhealthy individuals, women and men, a paired study was carried out: 40 unhealthy men with 40 unhealthy women, each of whom was matched with six healthy controls for age and sex (480 total). Finally, CPPQ-Mohedo showed a similar discriminant capacity between men and women. The dimensions involved (pain and quality of life) showed internal consistency, with Cronbach's alpha coefficient being 0.75.
Evaluation of the impact of pelvic floor dysfunction symptoms with the PFDI-20 (Pelvic Floor Distress Inventory) questionnaire | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  This questionnaire is the validated Spanish version of the Pelvic Floor Distress Inventory Short Form (PFDI-20). It is a reliable and valid instrument to assess symptoms and quality of life in Spanish women with pelvic floor dysfunction. The Spanish version achieved good semantic, conceptual, idiomatic, and content equivalence, with Cronbach's alpha coefficient being 0.837. This questionnaire has 20 items grouped into 3 components: Genital Prolapse Symptom Impact Questionnaire (POPDI, Cronbach's alpha= 0.787) with 6 items that assess symptoms of genital prolapse; Colorectal-Anal Symptom Impact Questionnaire (CRADI, Cronbach's alpha= 0.630) with 8 items that assess colorectal-anal symptoms; Urinary Symptom Impact Questionnaire (UDI, Cronbach's alpha= 0.699) with 6 items that assess urinary symptoms.
Assesment of menopausal symptoms with the Menopause Rating Scale (MSR). | The evaluation will be done at baseline before treatment and 6 weeks post treatment
  The Menopause Rating Scale (MRS) is a tool to assess the health-related quality of life of menopausal women. It is a standardized scale that meets psychometric standards, versioned in 9 languages. The scale was designed and standardized as a self-administered scale to (a) assess symptoms, (b) to assess the severity of symptoms over time, and (c) to measure changes before and after replacement therapy. menopause. It consists of 11 items (symptoms and complaints) evaluated from 0 (no complaint) to 4 (severe symptom). The degree of internal consistency (Cronbach's alpha coefficient) varies by country, ranging between 0.6 and 0.9.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín-Valero, PhD, Principal Investigator — University of Malaga
Locations (1):
- University of Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No